CLINICAL TRIAL: NCT06494488
Title: Differential Thrombogenesis Effects of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) Mediated by High-Density Lipoprotein (HDL)
Brief Title: Differential Thrombogenesis by EPA and DHA Mediated by HDL
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2133207; 7R01HL159204-02 (NIH)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lipid Metabolism Disorders; Hypertriglyceridemia
Keywords: Fish oil; Atherogenic lipidemia; Lipoproteins
MeSH Terms: conditions — Lipid Metabolism Disorders; Hypertriglyceridemia | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DHA group (Experimental): Participants will receive DHA supplement. 3 gelcaps, three times per day with meals (breakfast, lunch, and dinner). DHA supplement regimen contains 450 mg DHA and minimal EPA (60 mg) per pill.
  Participants will be given 28-day food and activity log.
  Interventions: Drug: DHA
- EPA group (Experimental): Participants will receive EPA supplement. 2 gelcaps, two times per day with meals (breakfast and dinner). 1 gelcap consists of 1 gram of EPA.
  Participants will be given 28-day food and activity log.
  Interventions: Drug: EPA

INTERVENTIONS:
Drug: EPA — Fish oil
  Other Names: eicosapentaenoic acid
  Arms: EPA group
Drug: DHA — Fish oil
  Other Names: docosahexaenoic Acid
  Arms: DHA group

SUMMARY:
The goal of this study is to learn more about omega-3 polyunsaturated fatty acids supplementation on blood lipid profile and platelets in patients with high cholesterol levels.

The purpose of this research is to gather information on the safety and effect of two different fish oils, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA).

Participants will:

Visit the clinic 3 times during study checkups, tests and blood collection. Randomized to either the EPA or the DHA supplementation group. Be given a 28-day food and activity log.

DETAILED DESCRIPTION:
Epidemiological studies suggest that consumption of omega-3 polyunsaturated fatty acids (n-3 PUFAs) derived from fish oil, mainly consisting of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), is associated with lower cardiovascular risk. However, interventional clinical trials aimed at reducing cardiovascular incidents by n-3 PUFAs supplementations have yielded inconsistent results. An intriguing fact is that only the outcome trials using EPA, but not those testing EPA/DHA mixed regimens, showed beneficial results. This discrepancy begs the question of whether EPA and DHA have differential effects and whether DHA blunts the cardiovascular benefits of EPA. However, no head-to-head clinical trial comparison of the biological effects of EPA and DHA in the hyperlipidemia patients has been reported. Hence, a well-designed, controlled, proof-of-concept clinical study testing EPA versus DHA in a relevant population is urgently required. In this study, the human subjects with atherogenic dyslipidemia will be randomized to dietary supplementation with four grams of either EPA or DHA n-3 PUFAs for eight weeks. At baseline and after the supplementation, various markers of thrombogenesis will be assessed, including biomarkers of the clotting cascade, thromboelastography, urinary thromboxane metabolites, whole blood aggregation, platelet aggregation, and flow cytometry analysis of platelets and platelet-leukocyte aggregates will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Fasting TG levels ≥ 150 mg/dL and < 500 mg/dL and HDL-C ≤ 40 (men) or ≤ 50 (women)
* LDL-C > 40 mg/dL and ≤ 130 mg/dL
* Able to provide informed consent and adhere to study schedules
* Agree to follow and maintain a relatively stable and low fatty fish intake diet (<3 servings per week)

Exclusion Criteria:

* Female with pregnancy, planned pregnancy (within the study period), or currently breastfeeding.
* Subjects with weight changes greater than 20% over the past 3 months
* Subjects planning a significant change in diet or exercise levels
* Malabsorption syndrome and/or chronic diarrhea
* Use of dietary supplements containing n-3 PUFA fatty acids
* Frequent consumption of n-3 PUFA-enriched fish (>3 times a week)
* Abnormal liver, kidney, or thyroid functions
* Drug or alcohol abuse within 6 months or significant mental/psychological impairment
* Current smokers
* Subjects taking daily aspirin, NSAIDs, anticoagulant, or corticosteroids
* Subjects with known bleeding disorders (for example, hemophilia)
* Known sensitivity or allergy to fish, shellfish, or omega-3 fatty acid supplements
* Subjects requiring regular transfusions for any reason
* No ethnic/racial groups will be excluded

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Platelet Aggregation Area Under the Curve (AUC) Over Time | 8 weeks
  Platelet aggregation will be assessed as the primary endpoint. The percentage of platelet aggregation will be measured at multiple time points, and the area under the curve (AUC) will be calculated to serve as a comprehensive marker of platelet aggregation response. Data will be presented as mean ± standard deviation or other appropriate statistical summaries.

SECONDARY OUTCOMES:
Percentage of Activated Platelets as Assessed by Flow Cytometry | 8 weeks
  Platelet activation will be assessed as a secondary endpoint. The percentage of activated platelets will be measured using flow cytometry, focusing on markers such as P-selectin expression and fibrinogen binding to the GPIIb/IIIa receptor. Measurements will be taken at multiple time points, and data will be summarized using statistical measures such as mean ± standard deviation.
Urinary Thromboxane Metabolite Levels normalized to urinary creatinine levels in ng/mmol | 8 weeks
  Urinary thromboxane metabolite levels will be measured as a secondary endpoint to evaluate thromboxane production. Quantification will be conducted using liquid chromatography-tandem mass spectrometry (LC-MS/MS). Results will be normalized to urinary creatinine levels (nanograms per millimole of creatinine) to account for variations in urine concentration. Data will be summarized using statistical measures such as mean ± standard deviation or other appropriate metrics.
Plasma levels of CRP in mg/L | 8 weeks
  Inflammatory markers will be measured as secondary endpoints to evaluate systemic inflammation. Plasma levels of C-reactive protein (CRP) will be reported in milligrams per liter (mg/L) using enzyme-linked immunosorbent assay (ELISA) or similar validated methods. Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma levels of resolvins in pg/mL | 8 weeks
  Specialized pro-resolving mediators (SPMs) will be measured as secondary endpoints to assess their role in inflammation resolution. Plasma levels of resolvins will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and reported in picograms per milliliter (pg/mL). Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma Levels of IL-6 in pg/mL | 8 weeks
  Inflammatory markers will be measured as secondary endpoints to evaluate systemic inflammation. Plasma levels of interleukin-6 (IL-6) will be quantified in picograms per milliliter (pg/mL) using enzyme-linked immunosorbent assay (ELISA) or similar validated methods. Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma Levels of TNF-α in pg/mL | 8 weeks
  Inflammatory markers will be measured as secondary endpoints to evaluate systemic inflammation. Plasma levels of tumor necrosis factor-alpha (TNF-α) will be quantified in picograms per milliliter (pg/mL) using enzyme-linked immunosorbent assay (ELISA) or similar validated methods. Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma levels of protectins in pg/mL | 8 weeks
  Specialized pro-resolving mediators (SPMs) will be measured as secondary endpoints to assess their role in inflammation resolution. Plasma levels of protectins will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and reported in picograms per milliliter (pg/mL). Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma levels of maresins in pg/mL | 8 weeks
  Specialized pro-resolving mediators (SPMs) will be measured as secondary endpoints to assess their role in inflammation resolution. Plasma levels of maresins, will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and reported in picograms per milliliter (pg/mL). Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.

CONTACTS AND LOCATIONS:
Overall Officials: Wenliang Song, MD, Principal Investigator — LIFESPAN CARDIOVASCULAR INSTITUTE
Locations (1):
- Brown University Health - Lipid Clinic, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No